CLINICAL TRIAL: NCT02862808
Title: Molecular Diagnosis of Syndromic or Isolated Severe Intellectual Disability Using Whole Exome Sequencing : a Pilot Study
Acronym: SHD-DI
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Other Study IDs: P/2015/242
Record Dates: First submitted 2016-08-08; First posted 2016-08-11 (Estimated); Last update posted 2020-07-22 (Actual); Status verified 2020-07

CONDITIONS: Severe Intellectual Disability
Keywords: Whole exome sequencing; Molecular diagnostic; Genetic counselling
MeSH Terms: conditions — Intellectual Disability

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Evaluation of diagnostic whole exome sequencing in patients with syndromic or isolated severe intellectual disability without a molecular diagnostic, with suspected autosomal recessive inheritance, allowing accurate genetic counseling in this high risk of recurrence group of diseases

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of syndromic or isolated severe intellectual disability (IQ <50) without a molecular diagnosis
* Recurrence in siblings (multiplex families) suggesting autosomal recessive inheritance (with or without parental consanguinity) or sporadic cases from a consanguineous union
* Conventional genetic tests performed (including array-CGH) and MRI/CT-scan available
* DNA samples from parents and from both unaffected or affected siblings available, for parental segregation and confirmation of candidate variations identified.
* Availability of a signed informed consent
* To be affiliated or beneficiary of French social security/healthcare system

Exclusion Criteria:

* Parents in the exclusion period of another study or as provided by the national register of volunteers
* High-probability diagnostic hypothesis for which a molecular test is available at lower cost than exome sequencing

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Retrospectively included patients presenting severe intellectual disability without a molecular diagnosis, born from consanguineous parents and / or with intra-familial recurrence, whose parents are requesting for molecular diagnosis, in a context of deadlock with conventional techniques
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2019-03-15 (Actual); Primary Completion 2019-12-03 (Actual); Study Completion 2019-12-03 (Actual)

PRIMARY OUTCOMES:
Number of patients with a molecular diagnostic and diagnostic yield | up to 12 months

SECONDARY OUTCOMES:
Cost/diagnostic ratio in comparison with conventional techniques | up to 12 months
Reporting time in comparison with conventional techniques | up to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Paul Kuentz, MD, Principal Investigator — Centre Hospitalier Universitaire de Besancon
Locations (1):
- CHU Besancon, Besançon, France

IPD SHARING:
Plan to Share IPD: No